CLINICAL TRIAL: NCT01864473
Title: Single Case Study of Vaginal Fistula Managed by Kshar Sutra, a Minimal Invasive Treatment.
Brief Title: Management of Vaginal Fistula by Kshar Sutra, a Minimally Invasive Treatment
Acronym: Bhagandar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government Ayurved College and Hospital (Other Government)
Responsible Party: Principal Investigator, Dr.Nita Mahadevrao Kedar, Associate professor, Government Ayurved College and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1234
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Vaginal Fistula
Keywords: Fistula , Bhagandar
MeSH Terms: conditions — Vaginal Fistula; Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Kshar Sutra (Other)
  Interventions: Other: Kshar Sutra

INTERVENTIONS:
Other: Kshar Sutra — The Kshar Sutra is a standard medicated thread smeared with Kshar of Apamarga (Achyranthus Aspera), Shnuhi (Euforbia Nerrifolia) which has quality of cutting and Haridra (Curcuma longa) which is used as a antiseptic. This combination of medicine on the thread helps in debridement and simultaneously healing of track. After conformation of vaginal fistula the track was cleaned with betadine and Hydrogen peroxide. The Kshar Sutra was tied covering the entire underlying track for simultaneous cutting and healing under all aseptic precaution. The patient was discharged on the next day of procedure. Patient was advice for Sitz bath with lukewarm water. The Kshar Sutra was changed weekly.
  Other Names: Medicated thread

SUMMARY:
Background:Fistula-in-ano is described as Bhagandara in the classics of Ayurveda, is an ancient surgical problem. It was commonly described even in the Vedic period. The description of Bhagandara, with the full text of its managements, can be gathered from the Sushruta Samhita, which is supposed to have been written in the second century B.C. Fistula-in-ano is a tubular ulcer formed around the peri-anal region. It may also be found anywhere in the perineal region. Its ramifications can extend to the lower back, subscrotal region, vagina etc.

Hypothesis:In Sushruta Samhita(2nd BC) Acharya Sushruta has advocated Kshar Sutra treatment due to probability of recurrence after surgery. The present treatment modality Kshar Sutra has been found effective and as adjuvant therapy by avoiding recurrence.

DETAILED DESCRIPTION:
A 42 years old female patient , come to the Shalyatantra O.P.D. of Government Ayurved Hospital,Nagpur with complaints of recurrent discharging boil at right side of Perianal region along with pain and discomfort in October 2010.

She gave a surgical history of incision and drainage for gluteal abscess done in year 2008 and after six month. The same complaint recurred after next six month .On local examination Patient had discharging sinus at 9 o clock position on right side of Perianal region. Before planning the treatment other etiologies like tuberculosis, diabetes mellitus , HIV or trauma were ruled out.

For the conformation of diagnosis Fistulogram was performed suggestive of low anal fistula with posterior internal opening. So under spinal anaesthesia probing was done. But it came to know that the track was directed upward in vagina and it had not any other opening in anal canal. Length of the tract was 7cm.

After conformation of vaginal fistula the track was cleaned with betadine and Hydrogen peroxide. The Kshar Sutra was tied covering the entire underlying track for simultaneous cutting and healing under all aseptic precaution. The patient was discharged on the next day of procedure. Patient was advice for Seitz bath with lukewarm water. The Kshar Sutra was changed weekly. To promote healing and to reduce pain and inflammation oral antibiotics, anti-inflammatory medicine were also prescribed.

The total period of Kshar Sutra treatment was two month. The track cut trough and simultaneously healed. It was observed that healing rate was slow as compare to cutting rate. In this patient. The patient was observed for a period of two year to check for recurrence.

The Kshar Sutra is a standard medicated thread smeared with Kshar of Apamarga (Achyranthus Aspera), Shnuhi (Euphorbia Nerrifolia)latex which has quality of cutting and Haridra (Curcuma Longa) which is used as a antiseptic. This combination of drugs on the thread helps in debridement and simultaneously healing.

ELIGIBILITY:
Inclusion Criteria:

* without any major illness like Diabetes, Hypertension, Asthma, Tuberculosis, and without multiple track.

Exclusion Criteria:

* with Major illness, multiple Fistulas, associated anorectal conditions

Ages: 42 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of Ksharstra in Vaginal Fistula | 1year
  Efficacy of Ksar Sutra in the management of Vaginal Fistula.

SECONDARY OUTCOMES:
Recurrence of Vaginal Fistula | 1year
  Efficacy of Kshar Sutra in Vaginal Fistula and its recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Nita M Kedar, M.S.(Ayu), Principal Investigator — Government Ayurved Hospital
Locations (1):
- Dr.Nita Mahadevrao Kedar, Nagpur, Maharashtra, India